CLINICAL TRIAL: NCT06791369
Title: The Prevalence of RYR1-related Disease - an International, Collaborative Multicentre Study
Brief Title: The Prevalence of RYR1-related Disease
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Radboud University Medical Center (Other); University of Leeds (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 335736
Record Dates: First submitted 2024-12-17; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Neuromuscular Disease; Malignant Hyperthermia; Congenital Myopathy; Multiminicore Disease; Nemaline Myopathy; Centronuclear Myopathy; Central Core Disease; Congenital Fiber Type Disproportion
Keywords: RYR1; Ryanodine Receptor Type 1; Malignant Hyperthermia; Congenital Myopathy
MeSH Terms: conditions — Neuromuscular Diseases; Malignant Hyperthermia; Myotonia Congenita; Minicore Myopathy with External Ophthalmoplegia; Myopathies, Nemaline; Myopathies, Structural, Congenital; Myopathy, Central Core

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biospecimens will not be collected. Pre-existing diagnostic data will be transferred by the direct clinical care team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The skeletal muscle ryanodine receptor (RYR1) gene encodes an important calcium channel in skeletal muscle, with an important role in muscle contraction. Mutations (i.e. disease-causing changes) in RYR1 are associated with an immensely wide range of clinical problems, ranging from inborn muscle conditions with profound weakness at birth ("congenital myopathies"), to a potentially fatal anaesthesia complication ("Malignant Hyperthermia, MH") in otherwise healthy individuals. Although RYR1-related conditions are believed to be amongst the most common neuromuscular disorders, their precise prevalence (i.e. the number of cases in a particular population at a given time) is currently unknown. Moreover, there is no information regarding the relative frequency of specific congenital myopathies, MH and related manifestations, such as the associated bleeding abnormality recently described by our team.

The lack of reliable prevalence data represents a major obstacle to addressing the needs of individuals affected by RYR1-related conditions, to appropriate resource allocation, and to preparation for clinical studies ("trial-readiness") essential for therapy development.

To address this shortcoming, we will conduct an international collaborative study involving neuromuscular and MH centres from the UK and the Netherlands, focusing on the prevalence of RYR1-related conditions, as a group and per subtype. The countries participating in this study were included because of 1) centralized RYR1 testing, 2) the presence of at least one database/registry with population-wide coverage capturing RYR1-related disorders and 3) of national myopathy and MH expertise centres. Information regarding RYR1-mutated individuals and their specific diagnosis will be obtained from national databases/registries, and analysed utilizing statistical methods that are well-established in the field of epidemiology.

This study will provide important information regarding the actual disease burden of RYR1-related disorders on a wider scale, inform appropriate research resource allocation, and preparation for trial readiness. This study will be funded by the RYR1-Foundation.

DETAILED DESCRIPTION:
ABSTRACT

The skeletal muscle ryanodine receptor (RYR1) gene encodes an important calcium channel in skeletal muscle, with a crucial role in muscle contraction. Mutations (i.e. disease-causing changes) in RYR1 are associated with a very wide range of clinical problems, ranging from inborn muscle conditions with profound weakness at birth ("congenital myopathies"), to a potentially fatal anaesthesia complication ("Malignant Hyperthermia, MH") in otherwise healthy individuals. Although RYR1-related conditions are believed to be amongst the most common neuromuscular disorders, their precise prevalence (i.e. the number of cases in a particular population at a given time) is currently unknown. Moreover, there is no information regarding the relative frequency of specific congenital myopathies, MH and related manifestations.

The lack of reliable epidemiological data represents a major obstacle to addressing the needs of individuals affected by RYR1-related conditions, to appropriate resource allocation, and to preparation for clinical studies ("trial-readiness") essential for therapy development. To address this shortcoming, we will conduct an international collaborative study involving neuromuscular and MH centres from the UK and the Netherlands, focussing on the prevalence of RYR1-related conditions, as a group and per subtype. The countries participating in this study were included because of 1) centralized RYR1 testing, 2) the presence of at least one database/registry with population-wide coverage capturing RYR1-related disorders and 3) of national myopathy and MH expertise centres. Information regarding RYR1-mutated individuals and their specific diagnosis will be obtained from national databases/registries, and analysed utilizing statistical approaches well-established in the epidemiological assessment of human disease and other mammalian populations.

This study will provide important information regarding the actual disease burden of RYR1-related disorders on a worldwide scale, inform appropriate research resource allocation, and preparation for trial readiness.

I. RYR1 RESEARCH PRIORITY AREA

A. Prevalence of RYR1-related Diseases

II. IMPACT ON RYR1-RELATED DISEASE

There are several reasons why this research is important and will make a significant difference in the RYR-1 Foundation's mission of finding treatments and cures for RYR1-related diseases:

For the first time, this study will provide reliable and up-to-data epidemiological data concerning the prevalence of RYR1-related disorders as a group, and with regards to specific subgroups within this wider group. Currently available epidemiological data are outdated and do not reflect the changes in diagnostic practices and the related increase in diagnostic yield over the last decade. Moreover, in contrast to the few currently available, regionally limited studies, this is the first epidemiological study concerning RYR1-related disorders taking a nationwide approach involving two large European countries with ethnically mixed populations, thus limiting the potential impact of regional differences in expertise and diagnostic rigour. Moreover, unlike previous studies this study will not only focus on RYR1-related myopathies but on RYR1-related disorders in their entirety, including congenital myopathies and malignant hyperthermia susceptibility.

Reliable epidemiological data concerning a group of disorders and/or specific subgroups within are an essential part of the preparation for clinical trial readiness, and will enable clinical translation of novel therapeutic developments concerning RYR1-related disorders into clinical practice. A number of novel therapeutic approaches are currently at the pre-clinical or clinical trial stage, with some of these approaches expected to be introduced into clinical practice over the next few years.

This study will highlight the true societal and individual disease burden of RYR1-related disorders and provide a stimulus for the appropriate allocation of health and research resources dedicated to this important group of neuromuscular disorders. Moreover, highlighting the relative frequency of specific subgroups (i.e. congenital myopathies, MH) within the wider group of RYR1-related disorders will help to focus and tailor future research efforts, as the underlying pathogenic mechanisms and individual disease manifestations in different subgroups are widely different. More importantly, therapeutic strategies aimed at patients suffering from congenital myopathies will not necessarily benefit those suffering from MH, and different treatment approaches based on reliable epidemiological data may be required.

Finally, obtaining more detailed genotype-phenotype data is likely to provide important insights in the currently not fully explored links between congenital myopathy and malignant hyperthermia phenotypes, and the intriguing continuum between malignant hyperthermia susceptibility, exertional myalgia/rhabdomyolysis and enhanced athletic performance, respectively.

III. SPECIFIC AIMS AND RATIONALE

The specific primary aims of this project are i) to investigate the prevalence of RYR1-related disorders in two different countries, the United Kingdom and the Netherlands; ii) to delineate the relative frequency of specific subgroups (in particular congenital myopathies vs Malignant Hyperthermia) within the overall group of RYR1-related disorders; and iii) to establish genotype-phenotype correlations for specific subgroups of RYR1-related myopathies and related disorders.

Although not a primary aim of this study, the designated Post-doctoral researcher will also be invited to contribute to other ongoing work on RYR1-related disorders from the department.

i) Prevalence of RYR1-related disorders: It is assumed that mutations in RYR1 are one of the most common genetic causes of non-dystrophic neuromuscular disorders, however, there are currently only few studies reporting the prevalence of these common conditions. Moreover, these studies are regionally limited and more than 10 years old, not reflecting recent changes and regional differences in diagnostic practice. An international collaborative study focussing on the prevalence of RYR1-related disorders is therefore much needed and timely.

ii) Frequency of specific subgroups of RYR1-related disease: Over the last two decades, the spectrum of RYR1-related disorders has continuously evolved, encompassing a very wide range of conditions, including several congenital myopathies (in particular, Central Core Disease, CCD; Multi-minicore Myopathy, MmD; Centronuclear Myopathy, CNM; Congenital Fibre Type Disproportion, CFTD), Malignant Hyperthermia Susceptibility (MHS), and related permanent (King-Denborough Syndrome, KDS) and episodic (exertional rhabdomyolysis, ERM; atypical periodic paralysis) myopathies. There are currently no data regarding the frequency of these specific subgroups, and a specific study addressing this shortcoming is urgently needed.

iii) Genotype-phenotype correlations in RYR1-related disorders: Defining genotype-phenotype correlations will help to further elucidate the complex relationship between RYR1-related MHS and CM phenotypes, and provide the basis for future research, including functional studies. Specific analyses to be undertaken will, for example, focus on RYR1 variants implicated in King-Denborough syndrome (KDS), a rare myopathy associated with dysmorphic features and profound malignant hyperthermia susceptibility (MHS), and on the p.Thr4288_Ala4290dup, a RYR1 variant found at detectable frequency in individuals of African ancestry on databases of genomic variation, often associated with increased athletic ability. RYR1 p.Thr4288_Ala4290dup has also been found in individuals with exertional myalgia/rhabdomyolysis (ERM) and malignant hyperthermia (MH), but it is currently unclear if this observation reflects a causal association or just the relatively high frequency of this variant in certain populations. To resolve this question, we will compare the frequency of p.Thr4288_Ala4290dup in the datasets obtained in i) and ii) with its population frequency.

IV. PRELIMINARY/SUPPORTING DATA

i) Prevalence of RYR1-related disorders: There is currently only one study from the United States, indicating the prevalence of RYR1-related congenital myopathies as 1 in 90000 in a representative Paediatric population (Amburgey et al., Ann Neurol 2011;70:662-665); this is likely to be an underestimate, considering that this more than 10-year-old study precedes the widespread introduction of next generation sequencing into clinical diagnostics, and does not take into account presentations such as MH, or MH-related manifestations (such as exertional myalgia/rhabdomyolysis and late-onset axial myopathy) that have only been recognized over the last decade. A more recent UK-based study indicates mutations in RYR1 as the most common identifiable genetic cause of congenital myopathies [Maggi et al., Neurology 2015;84:28-35], but does not comment on their overall prevalence.

ii) Frequency of specific subgroups of RYR1-related disease: There is currently only one study from the UK concerning the frequency of specific RYR1-related congenital myopathies (CMs), suggesting that Central Core Disease (CCD) and Multi-minicore Disease (MmD) (the "core myopathies") are most common, whilst others such as Centronuclear Myopathy (CNM) and Congenital Fibre Type Disproportion (CFTD) are less frequent [Maggi et al., Neurology 2015;84:28-35]. There is currently no information regarding the relative frequency of CM versus malignant hyperthermia phenotypes, and of more recently emerged MH-associated manifestations such as exertional myalgia/rhabdomyolysis and late-onset axial myopathy.

iii) Genotype-phenotype correlations in RYR1-related disorders: Defining genotype-phenotype correlations will help to further elucidate the complex relationship between RYR1-related MHS and CM phenotypes, and provide the basis for future research, including functional studies. Specific analyses to be undertaken will, for example, focus on RYR1 variants implicated in King-Denborough syndrome (KDS), a rare myopathy associated with dysmorphic features and profound malignant hyperthermia susceptibility (MHS), and on the p.Thr4288_Ala4290dup, a RYR1 variant found at detectable frequency in individuals of African ancestry on databases of genomic variation, often associated with increased athletic ability. RYR1 has also been found in individuals with exertional myalgia/rhabdomyolysis (ERM) and malignant hyperthermia (MH), but it is currently unclear if this observation reflects a causal association or just the relatively high frequency of this variant in certain populations. To resolve this question, we will compare the frequency of p.Thr4288_Ala4290dup in the datasets obtained in i) and ii) with its population frequency.

V. DETAILED PROJECT DESCRIPTION

1) EXPERIMENTAL PLAN AND METHODS:

A) Study description:

i) Prevalence of RYR1-related disorders: To determine the prevalence of RYR1-related disorders, we will collect demographic, genetic, clinical and pathological data from patients diagnosed and reviewed in two different countries, the United Kingdom and the Netherlands, with populations of 67 and 17 million, respectively. Above countries will be included based on the availability of a) centralized RYR1 testing with population-wide coverage, and/or the presence of national expertise centres for b) congenital myopathies and malignant hyperthermia (MH) with patient databases/registries with population-wide coverage.

Inclusion criteria for patients are a) the presence of (an) unequivocally pathogenic RYR1 mutation(s), b) clinical features of a recognized RYR1-related disorder (i.e. a congenital myopathy, MH or related phenotypes), c) at least one specialist review at one of the national expertise centres and d) being resident in one of the participating countries. Criteria for the diagnosis of a congenital myopathy are the presence of suggestive clinical features and supportive muscle biopsy findings, or the presence of supportive histopathological findings in a first degree relative with similar clinical features and the same RYR1 genotype. Criteria for the diagnosis of MH susceptibility are clinical features suggestive of malignant hyperthermia (as defined by a diagnostic Larach score) and/or a positive IVCT/CHCT test, or a relative with a history of MH and the same RYR1 genotype. Exclusion criteria will be a clinical diagnosis of a congenital myopathy or malignant hyperthermia without any of the supportive evidence as outlined above, or not being resident in one of the participating countries.

Data collection: For each patient, we will collect the following data from databases/registries already existing at the participating centres: Age at diagnosis, sex and RYR1 genotype. We will also collect details regarding the specific RYR1-related diagnosis, categorized as Central Core Disease (CCD), Multi-minicore Disease (MmD), Centronuclear Myopathy (CNM), Congenital Fibre Type Disproportion (CFTD), King-Denborough Syndrome (KDS), congenital myopathy with non-specific histopathological features (CMNS), Malignant Hyperthermia Susceptibility (MHS) and Exertional Rhabdomyolysis/Myalgia (ERM). In cases with more than one diagnosis of a RYR1-related disorders (for example, CCD and MH), both diagnoses will be recorded. Data will be collected for all patients fulfilling the inclusion criteria seen at one of the participating centres over a 10-year period, between 01.01.2011 to 31.12.20. All data will be stored in anonymized form on a secure server at King's College University, London. A standardized data collection proforma has been discussed and agreed will be provided separately.

Statistical and epidemiological analysis: Point prevalences for each country will be calculated based on the number of patients alive on the 31.12.2020, in comparison to national population numbers. In countries where more than one population-based database/registry capturing RYR1-related disorders is available, we will also perform a multiple source capture-recapture approach (as described in detail by Deenen et al.,Neurology 2014;83:1056-59), an approach suitable to correct for symptomatic individuals that may not have been captured in any of the interrogated databases/registries. The rates will be calculated in the annual cohorts for the observation period, and will be expressed per 100,000 persons per year. Rates will presented for the overall cohort and specified subgroups, each stratified by age and sex. All incidences will be age-adjusted using direct methods to the 2013 European Standard Population. The 95% CIs will be estimated assuming a Poisson distribution for the number of events.

ii) Frequency of specific subgroups of RYR1-related disease: Based on the data obtained in i), we will also calculate the frequency of specific subgroups of RYR1-related disorders, including the various congenital myopathies (CCD, MmD, CNM, CFTD, CMNS) and Malignant Hyperthermia (MH). For each patient, the clinical and histopathological diagnosis will be verified by review of the clinical notes and the original muscle biopsy wherever possible.

iii) Genotype-phenotype correlations in RYR1-related disorders: We have previously published the largest series of RYR1-related KDS patients so far, indicating that KDS is a unique myopathy closely linked to MH-associated RYR1 mutations, but with the precise mode of inheritance currently unresolved [Dowling et al., Neuromuscul Disord 2011;21:420-427]. We have subsequently identified more than 10 additional patients with RYR1-related KDS and found an apparent association with the RYR1 central domain MH mutational hotspot (Fernandez-Garcia et al., manuscript in preparation), an observation that needs to be validated in larger datasets.

The RYR1 p.Thr4288_Ala4290dup has been previously reported in association with MH reactions, often in individuals carrying at least one additional RYR1 variant [Levano et al., Hum Mutat 2008;30:590-8; Sambuughin et al., Clin Genet 2009;76:564-68]. We have also found RYR1 p.Thr4288_Ala4290dup in a cohort of patients presenting with RYR1-associated exertional myalgia/rhabdomyolysis, often associated with an apparently enhanced athletic ability [Dlamini et al. Neuromuscul Disord 2013;23:540-48], an association that has not yet been explored further.

B) Ethical considerations, regulatory requirements and data management protocol:

The study has received preliminary Research Ethics Committee (REC) approval by the King's College London REC pending some minor amendments (KCL Ethics Ref: LRS/DP-22/23-36029).

A data management protocol has been developed by the designated data manager for the study. The retrospective data collected from the United Kingdom (Guy's & St Thomas' NHS Foundation Trust, London, Great Ormond Street Children's Hospital, London and the National Malignant Hyperthermia Centre, Leeds), and the Netherlands (Radboud University Medical Centre, Nijmegen) will not have any direct patient identifiers or any patient pseudonyms that allows patient re-identification. The data from these centres will by anonymised. Data collected will be for as much as 1000 patients and transferred from each centre through a secured encrypted method, such as encrypted email depending on the size of the document being transferred. A data sharing agreement will be made with each centre detailing the data items to be shared, that data will be anonymised, and the mode of transfer. There will be no data transfer out from the study centre (Kings College London, KCL) to third parties. The study will run for two years, and its data will be retained and archived in compliance with the KCL Data Retention Schedule for 10 years. Through the KCL REMAS (Research Ethics Management Application System) the study will be registered with KDPR (King's Data Protection Register) in compliance with the UK Data Protection Act 2018.

ELIGIBILITY:
Inclusion Criteria:

* the presence of (an) unequivocally pathogenic RYR1 mutation(s)
* clinical features of a recognized RYR1-related disorder (i.e. a congenital myopathy, MH or related phenotypes)
* at least one specialist review at one of the national expertise centres
* being resident in one of the participating countries.

Criteria for the diagnosis of a congenital myopathy are the presence of suggestive clinical features and supportive muscle biopsy findings, or the presence of supportive histopathological findings in a first degree relative with similar clinical features and the same RYR1 genotype. Criteria for the diagnosis of MH susceptibility are clinical features suggestive of malignant hyperthermia (as defined by a diagnostic Larach score) and/or a positive IVCT/CHCT test, or a relative with a history of MH and the same RYR1 genotype. Exclusion criteria will be a clinical diagnosis of a congenital myopathy or malignant hyperthermia without any of the supportive evidence as outlined above, or not being resident in one of the participating countries.

Exclusion Criteria:

* a clinical diagnosis of a congenital myopathy or malignant hyperthermia without any of the supportive evidence as outlined above
* not being resident in one of the participating countries.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will collect the data from local databases/registries already existing at the participating centres:
  * Malignant Hyperthermia Investigation Unit, St James's University Hospital, Leeds
  * Great Ormond Street Hospital, London
  * Evelina London Children's Hospital, London
  * Radboud University Medical Centre, Nijmegen
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The prevalence of RYR1-related disorders | Jan 2011 - Dec 2020
  To determine the prevalence of RYR1-related disorders, we will collect demographic, genetic, clinical and pathological data from patients diagnosed and reviewed in two different countries, the United Kingdom and the Netherlands, with populations of 67 and 17 million, respectively.
  Point prevalences for each country will be calculated based on the number of patients alive on the 31.12.2020, in comparison to national population numbers.

SECONDARY OUTCOMES:
Determine frequency of subgroups of RYR1-related disorders | Jan 2011 - Dec 2020
  Based on the data obtained for the primary aim, we will also calculate the frequency of specific subgroups of RYR1-related disorders, including the various congenital myopathies (CCD, MmD, CNM, CFTD, CMNS) and Malignant Hyperthermia (MH). For each patient, the clinical and histopathological diagnosis will be verified by review of the clinical notes and the original muscle biopsy wherever possible.
To establish genotype-phenotype correlations in RYR1-related disorders | Jan 2011 - Dec 2020
  We will validate the apparent association between RYR1-related KDS and a RYR1 central domain MH mutational hotspot.
  The RYR1 p.Thr4288_Ala4290dup has been previously reported in association with MH reactions, often in individuals carrying at least one additional RYR1 variant [Levano et al., 2008; Sambuughin et al., 2009]. We have also found RYR1 p.Thr4288_Ala4290dup in a cohort of patients presenting with RYR1-associated exertional myalgia/rhabdomyolysis, often associated with an apparent enhanced athletic ability [Dlamini et al. 2013]; these associations will be validated in this larger dataset.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The decision not to share IPD is based on the sensitive nature of the data involved, which includes genetic information. Sharing genetic data carries inherent privacy and confidentiality risks, even with de-identification measures in place. Protecting the privacy of participants and complying with ethical standards and regulatory requirements are of utmost importance. Additionally, the potential for re-identification of individuals from genetic data presents a significant concern, which we aim to mitigate by restricting access.

REFERENCES:
- [Background] Zhou H, Lillis S, Loy RE, Ghassemi F, Rose MR, Norwood F, Mills K, Al-Sarraj S, Lane RJ, Feng L, Matthews E, Sewry CA, Abbs S, Buk S, Hanna M, Treves S, Dirksen RT, Meissner G, Muntoni F, Jungbluth H. Multi-minicore disease and atypical periodic paralysis associated with novel mutations in the skeletal muscle ryanodine receptor (RYR1) gene. Neuromuscul Disord. 2010 Mar;20(3):166-73. doi: 10.1016/j.nmd.2009.12.005. Epub 2010 Jan 18. PMID 20080402
- [Background] Wilmshurst JM, Lillis S, Zhou H, Pillay K, Henderson H, Kress W, Muller CR, Ndondo A, Cloke V, Cullup T, Bertini E, Boennemann C, Straub V, Quinlivan R, Dowling JJ, Al-Sarraj S, Treves S, Abbs S, Manzur AY, Sewry CA, Muntoni F, Jungbluth H. RYR1 mutations are a common cause of congenital myopathies with central nuclei. Ann Neurol. 2010 Nov;68(5):717-26. doi: 10.1002/ana.22119. PMID 20839240
- [Background] Maggi L, Scoto M, Cirak S, Robb SA, Klein A, Lillis S, Cullup T, Feng L, Manzur AY, Sewry CA, Abbs S, Jungbluth H, Muntoni F. Congenital myopathies--clinical features and frequency of individual subtypes diagnosed over a 5-year period in the United Kingdom. Neuromuscul Disord. 2013 Mar;23(3):195-205. doi: 10.1016/j.nmd.2013.01.004. Epub 2013 Feb 8. PMID 23394784
- [Background] Loseth S, Voermans NC, Torbergsen T, Lillis S, Jonsrud C, Lindal S, Kamsteeg EJ, Lammens M, Broman M, Dekomien G, Maddison P, Muntoni F, Sewry C, Radunovic A, de Visser M, Straub V, van Engelen B, Jungbluth H. A novel late-onset axial myopathy associated with mutations in the skeletal muscle ryanodine receptor (RYR1) gene. J Neurol. 2013 Jun;260(6):1504-10. doi: 10.1007/s00415-012-6817-7. Epub 2013 Jan 18. PMID 23329375
- [Background] Lopez RJ, Byrne S, Vukcevic M, Sekulic-Jablanovic M, Xu L, Brink M, Alamelu J, Voermans N, Snoeck M, Clement E, Muntoni F, Zhou H, Radunovic A, Mohammed S, Wraige E, Zorzato F, Treves S, Jungbluth H. An RYR1 mutation associated with malignant hyperthermia is also associated with bleeding abnormalities. Sci Signal. 2016 Jul 5;9(435):ra68. doi: 10.1126/scisignal.aad9813. PMID 27382027
- [Background] Levano S, Vukcevic M, Singer M, Matter A, Treves S, Urwyler A, Girard T. Increasing the number of diagnostic mutations in malignant hyperthermia. Hum Mutat. 2009 Apr;30(4):590-8. doi: 10.1002/humu.20878. PMID 19191329
- [Background] Jungbluth H, Zhou H, Hartley L, Halliger-Keller B, Messina S, Longman C, Brockington M, Robb SA, Straub V, Voit T, Swash M, Ferreiro A, Bydder G, Sewry CA, Muller C, Muntoni F. Minicore myopathy with ophthalmoplegia caused by mutations in the ryanodine receptor type 1 gene. Neurology. 2005 Dec 27;65(12):1930-5. doi: 10.1212/01.wnl.0000188870.37076.f2. PMID 16380615
- [Background] Dowling JJ, Lillis S, Amburgey K, Zhou H, Al-Sarraj S, Buk SJ, Wraige E, Chow G, Abbs S, Leber S, Lachlan K, Baralle D, Taylor A, Sewry C, Muntoni F, Jungbluth H. King-Denborough syndrome with and without mutations in the skeletal muscle ryanodine receptor (RYR1) gene. Neuromuscul Disord. 2011 Jun;21(6):420-7. doi: 10.1016/j.nmd.2011.03.006. Epub 2011 Apr 22. PMID 21514828
- [Background] Dlamini N, Voermans NC, Lillis S, Stewart K, Kamsteeg EJ, Drost G, Quinlivan R, Snoeck M, Norwood F, Radunovic A, Straub V, Roberts M, Vrancken AF, van der Pol WL, de Coo RI, Manzur AY, Yau S, Abbs S, King A, Lammens M, Hopkins PM, Mohammed S, Treves S, Muntoni F, Wraige E, Davis MR, van Engelen B, Jungbluth H. Mutations in RYR1 are a common cause of exertional myalgia and rhabdomyolysis. Neuromuscul Disord. 2013 Jul;23(7):540-8. doi: 10.1016/j.nmd.2013.03.008. Epub 2013 Apr 28. PMID 23628358
- [Background] Amburgey K, McNamara N, Bennett LR, McCormick ME, Acsadi G, Dowling JJ. Prevalence of congenital myopathies in a representative pediatric united states population. Ann Neurol. 2011 Oct;70(4):662-5. doi: 10.1002/ana.22510. PMID 22028225